CLINICAL TRIAL: NCT00659997
Title: Longitudinal Study of Efficacy of Standard Albendazole Treatment Versus Levamisole/Pyrantel Pamoate on Soil Transmitted Helminth Infections
Brief Title: Efficacy Albendazole and Levamisole Against STH on Unguja
Acronym: ALBvLEV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Natural History Museum, United Kingdom (Other Government)
Collaborators: Ministry of Health, Tanzania (Other Government); University of London (Other)
Responsible Party: Prof D Rollinson, Natural History Museum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHMDEWORMING
Record Dates: First submitted 2008-04-10; First posted 2008-04-17 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Ascariasis; Trichuriasis
Keywords: Ascariasis; Trichuriasis; Drug resistance
MeSH Terms: conditions — Ascariasis; Trichuriasis | interventions — Albendazole; Levamisole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 1 Individuals treated with Albendazole
  Interventions: Drug: Albendazole
- 2 (Active Comparator): Individuals treated with Levamisole
  Interventions: Drug: Levamisole

INTERVENTIONS:
Drug: Albendazole — Single oral dose of 400mg
  Arms: 1
Drug: Levamisole — Single oral dose of 2.5mg/kg
  Arms: 2

SUMMARY:
Field epidemiological studies undertaken during 2005 in four village locations in Northern Unguja, Zanzibar examined mothers and their pre-school aged children for helminth infections.

The prevalence of Ascaris lumbricoides was found to have remained relatively high despite community-wide treatment with the mass administration of Albendazole (a WHO recommended de-wormer) in coordination with community vitamin A supplementation.

One hypothesis for this is that the children and mothers had Ascaris infections more tolerant to Albendazole that subsequently failed to clear. It is necessary to compare the present drug efficiency of Albendazole (first-line de-wormer) with Levamisole (second-line de-wormer) on STH infections such patients a case-control setting to shed light on the putative resistance of local Ascaris/Trichuris to albendazole.

In so doing, this should clarify whether there is resistance developing towards Albendazole and have possible implications for introducing combination therapies of Levamisole and Albendazole for first line de-worming mothers and their children in the future.

DETAILED DESCRIPTION:
The study was conducted in 10 villages on Unguja Island representative of urban, semi-urban and rural environments. After liaison with the local Shehia (the elected community leader) mothers and their children aged between 6 months and 5 years old were invited to attend a walk-in mobile clinic. In accordance with WHO sample size recommendations of 30 individuals per site and to cater for drop-out/non-compliance, target enrolment was about 50 mother and child pairs at each study village.

Stool specimens were transported to the Helmtin Control Laboratory Unguja laboratory for visual inspection of stool consistency and presence of blood, after which a single Kato-Katz thick smear (41.7mg) was prepared. Eggs of all STH species were counted by inspection at 100x microscopy and expressed as a tally of eggs per gram (EPG). To ensure consistency of egg counts, slides were read by the same two technicians for each study village.

10 Mother and child pairs found positive for Ascaris and/or Trichuris were randomised, by coin tossing, to receive either a single tablet of ALB (400mg) or an appropriate dose of LEV (2.5 mg/kg). A parasitological follow-up took place 18 days after treatment where a requested stool sample was analyzed by a single Kato-Katz thick smear for assessment of STH clearance. In accordance with WHO's 'no survey without service' all attendees were given an additional ALB tablet.

ELIGIBILITY:
Inclusion Criteria:

* Presently with soil-transmitted helminthiasis

Exclusion Criteria:

* absence of soil-transmitted helminthiasis

Ages: 1 Year to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2006-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Clearance of STH faecal eggs in patient stool | 18 days

CONTACTS AND LOCATIONS:
Locations (1):
- Helminth Control Laboratory Unguja, Stone Town, Tanzania

REFERENCES:
- [Result] Stothard JR, Imison E, French MD, Sousa-Figueiredo JC, Khamis IS, Rollinson D. Soil-transmitted helminthiasis among mothers and their pre-school children on Unguja Island, Zanzibar with emphasis upon ascariasis. Parasitology. 2008 Oct;135(12):1447-55. doi: 10.1017/S0031182008004836. Epub 2008 Sep 8. PMID 18775092